CLINICAL TRIAL: NCT04740242
Title: ALCALOTIC Study: Metabolic Alcalosis in Decompensated Heart Failure: Prevalence and Influence on Prognosis
Brief Title: Metabolic Alkalosis in Heart Failure
Status: Completed | Type: Observational
Sponsor: Spanish Society of Internal Medicine (Other)
Responsible Party: Principal Investigator, Joan Carles Trullas Vila, Principal Investigator. Heart Failure Workin Group. Spanish Society of Internal Medicine, Spanish Society of Internal Medicine
Other Study IDs: ALCALOTIC
Record Dates: First submitted 2021-01-30; First posted 2021-02-05 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure; Metabolic Alkalosis; Diuretics Drug Reactions; Decompensated Heart Failure; Acute Heart Failure
Keywords: metabolic alkasosis; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort of exposed patients (Group 1): All patients admitted for decompensated HF and presenting MA at the time of admission
- Cohort of unexposed patients (Group 2): All patients admitted for decompensated HF and who do NOT present MA at the time of admission

SUMMARY:
Metabolic alkalosis (MA) is the most common acid-base disorder and when it's severe it can have effects on cellular function and contribute to an increase in mortality.

MA is a common complication of heart failure (HF) especially when patients are treated with diuretics, but few studies have analyzed the prevalence of acid-base disorders in patients with HF.

All these studies have shown that MA is more common in patients with HF in more advanced stages and that the use of diuretics increases the prevalence of MA.

The study hypothesis, based on clinical experience and the few data that exist in the scientific literature, is that MA is a frequent analytical disorder in patients admitted for decompensated HF and that its presence entails a worse short-term vital prognosis.

The ALCALOTIC study is an observational cohort and prospective study.

The main objectives of the study are the following:

1. To determine the prevalence of MA in patients admitted for decompensated HF
2. To analyze if there are differences in patients admitted for HF according to the presence of MA on admission
3. To determine if the presence of MA has an influence on the short-term prognosis in patients admitted for decompensated HF

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for decompensated HF (main admission diagnosis), who meet the diagnostic criteria of the 2016 European HF Guidelines and who sign the informed consent to participate in the study
* Patients must give their written consent to participate in the study

Exclusion Criteria:

* Patients whose main reason for admission is not decompensated HF. Those patients who are admitted for another reason and who also have decompensated HF secondarily cannot be included
* Patients who do not strictly meet the diagnostic criteria for HF of the European HF Guidelines.
* Patients for whom analytical values are not available in relation to acid-base balance at the time of admission
* Patients with a pathological history that can clearly justify metabolic alkalosis, such as primary or secondary hyperaldosterism
* Patients who were taking sodium bicarbonate prior to admission
* Patients with factors present at admission that may justify the presence of metabolis alkalosis: vomiting, diarrea, etc.
* Patients who do not give their consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from the Internal Medicine Services of Spanish Hospitals whose researchers are active members of the Working Group on Heart Failure and Atrial Fibrillation of the Spanish Society of Internal Medicine
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | an average of 7 days
  In-hospital mortality from all causes

SECONDARY OUTCOMES:
Mortality during follow-up | Mortality at 30 and 90 days after hospital discharge
  All-cause mortality 30 and 90 days after hospital discharge
Re-admission (all cause) during follow-up | Re-admission at 30 and 90 days after hospital discharge
  Re-admission for all causes 30 and 90 days after hospital discharge
Readmission for heart failure during follow-up | Readmission for heart failure 30 and 90 days after hospital discharge
  Re-admission for heart failure 30 and 90 days after hospital discharge
Lenght of Hospital stay | Lenght of Hospital stay will be determined the day of hospital discharge, an average of 7 days after admission/inclusion
  Lenght of Hospital stay during hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Service, Hospital d'Olot (Girona), Olot, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galla JH. Metabolic alkalosis. J Am Soc Nephrol. 2000 Feb;11(2):369-375. doi: 10.1681/ASN.V112369. No abstract available. PMID 10665945
- [Background] Peixoto AJ, Alpern RJ. Treatment of severe metabolic alkalosis in a patient with congestive heart failure. Am J Kidney Dis. 2013 May;61(5):822-7. doi: 10.1053/j.ajkd.2012.10.028. Epub 2013 Mar 5. PMID 23481366